CLINICAL TRIAL: NCT04891159
Title: Training in Shared Decision-making of Cystic Fibrosis Centers Competences in the Treatment of CF Related Diabetes in Adult Patients: a Qualitative Evaluation of the Implementation
Brief Title: Training in Shared Decision-making of Cystic Fibrosis Centers Competences in the Treatment of CF Related Diabetes in Adult Patients
Acronym: FORAIDMUCO
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL21_0085
Record Dates: First submitted 2021-04-16; First posted 2021-05-18 (Actual); Last update posted 2021-05-18 (Actual); Status verified 2021-03

CONDITIONS: Diabetes; Cystic Fibrosis
Keywords: Cystic Fibrosis; Shared decision-making; Treatments of diabete
MeSH Terms: conditions — Diabetes Mellitus; Cystic Fibrosis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Shared decision making: During the first consultation (V1), the doctor will present the patient on the therapeutic treatment information related to diabetes according to the shared decision making (options, benefits, risks) with the assistance of decision support tools. The decision-making visit will take place after a reflection period of 8 to 15 days after V1. A discussion based on the feedback from this period of reflection will take place between the two actors and either there is a common agreement on the decision taken (shared decision-making), or the decision is taken by the patient, or the decision is made by the physician at the request of the patient. A social sciences and humanities methodologist will attend each consultation, onsite or in videoconferencing. After the consultation, he realized a semi-structured interview with the patient. During this interview, the patient filled the self-administered questionnaires: SDM-Q-9, SURE, CollaboRATE, Spielberger test and the research team questionnaire
  Interventions: Other: Shared decision making
- Control group: Decision-making for insulin therapy is based on the usual practice defined in each Cystic Fibrosis Centers Competences with decision-making procedures specific to each center and doctor. The decision-making process is generally carried out in two consultations.
  A social sciences and humanities methodologist will attend each consultation, onsite or in videoconferencing.
  After the consultation, he realized a semi-structured interview with the patient. During this interview, the patient filled the self-administered questionnaires (SDM-Q-9, SURE, CollaboRATE, Spielberger test and the research team questionnaire).

INTERVENTIONS:
Other: Shared decision making — The intervention consists of 5 components: 1) Online shared decision making training (2 hours, e-learning); 2) Individual coaching for doctors by a shared decision making expert; 3) Implementation of the shared decision making; 4) Link to institutional approaches to patient engagement; 5) Integration of the shared decision making into the multidisciplinary consultation meetings of the Cystic Fibrosis Centers Competences.
  Groups: Shared decision making

SUMMARY:
Diabetes affects half of cystic fibrosis patients aged 30 years and older. It develops asymptomatically for a long time. Also, two options are possible: start insulin treatment now with the additional constraints associated with cystic fibrosis or wait while monitoring the patient's clinical status and initiate insulin treatment when he has developed symptoms and therefore later. In practice, the choice between these two options takes place over two medical consultations without a formalized shared decision-making process between the doctor and the patient.

Shared decision-making is a decision-making process in which the healthcare provider and the patient learn about patients care options and then deliberate to reach a common agreement on the decision taken.

Shared decision-making seemed particularly relevant to us in cystic fibrosis where there are complex treatment options with variable short-, medium- and long-term side effects and where the disease and its treatments have a high impact on the patient's quality of life.

ELIGIBILITY:
Inclusion Criteria:

Concerning the patient :

* Patient major
* Patient affected by cystic fibrosis
* Patient able to understand french
* Patient sable on Respiratory and nutritional status
* Patient with disorders of carbohydrate metabolism in the glucose tolerance test (OGTT)
* Patient with normal fasting blood sugar

Concerning the health professionals :

Medical and paramedical professionals practising in the adult Cystic Fibrosis Centers Competences (doctors, nurses, dieticians, psychologists, physiotherapists, etc...)

Exclusion Criteria:

* Patient with transplant
* Patient who have received insulin therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Major cystic fibrosis patients
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2021-09 (Estimated); Primary Completion 2023-04 (Estimated); Study Completion 2023-04 (Estimated)

PRIMARY OUTCOMES:
Adoption of a shared decision making measured by the total score obtained on the 9 items of the shared decision making questionnaire (SDM-Q-9), translated into French. | The principal endpoint is measured for interventional group : immediately after the second consultation, for control group : immediately after the consultation where the treatment decision is taken (consultation 1 or 2)
  The SDM-Q-9 is a self-administered questionnaire of 9 items coded on a 6-point Likert scale. A total score between 0 and 45 is calculated from the sum of the scores obtained for the 9 questions. This score is converted between 0 and 100 by multiplying by a factor of 20/9, 0 indicating a non adoption of shared decision making as perceived by the patient and conversely 100 indicating an adoption of shared decision making as perceived by the patient. The total score will be described in each group by mean, standard deviation, median, quartiles and extent, and will be compared between the 2 groups with a non-parametric Wilcoxon test.

CONTACTS AND LOCATIONS:
Locations (4):
- France (4):
  - CRCM Grenoble adulte - Hôpital Albert Michallon, La Tronche
  - CRCM Montpellier Mixte - Hôpital Arnaud de Villeneuve, Montpellier
  - CRCM Lyon adulte - Centre hospitalier Lyon Sud, Pierre-Bénite
  - CRCM Rennes adulte - Hôpital Pontchaillou, Rennes

REFERENCES:
- [Derived] Moumjid N, Gotte C, Hommey S, Poupon Bourdy S, Haesebaert J, Durieu I, Reynaud Q. Mixed Comparative Evaluation of a Training Program Dedicated to Cystic Fibrosis Reference Centers: Protocol for the Pilot Implementation of Shared Decision-Making in the Treatment of Diabetes in Adult Patients With Cystic Fibrosis. JMIR Res Protoc. 2025 Jan 28;14:e62931. doi: 10.2196/62931. PMID 39874570